CLINICAL TRIAL: NCT02647684
Title: Triple P for Parents of Children With a Diagnosis of Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: Royal Children's Hospital (Other)
Responsible Party: Principal Investigator, Katie Swift, Chief Investigaor, University of Manchester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 163356/15EM/0101
Record Dates: First submitted 2015-09-23; First posted 2016-01-06 (Estimated); Last update posted 2016-10-25 (Estimated); Status verified 2016-10

CONDITIONS: Cancer
Keywords: Cancer; Parenting; Self-directed Triple P
MeSH Terms: conditions — Neoplasms | interventions — (tris(diphenylphosphinomethyl)phenylborate)(p-tolylnitrido)iron(I)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Self- Direced Triple P (Experimental): Self-directed Triple P workbook to be completed over 10 weeks. Over the course of the workbook parents will think about the changes they would like to make to their child's behaviour. They are taught strategies to enhance their relationship with their child, and promote desirable behaviours. They learn about options for managing problem behaviours and have the opportunity to decide if they would like to use any of these approaches with their child in a clear and consistent way. Parents have practice period to use the approaches they have learnt in weeks 1-3. By the end of week 6 they will have had practice in using their chosen positive parenting approaches, learnt to set goals and monitor their own behaviour when using these strategies. The final weeks aim to help parents identify times when the strategies may not be working and provide survival tips on what to do at these times.
  Interventions: Behavioral: Self-Directed Triple P

INTERVENTIONS:
Behavioral: Self-Directed Triple P — 10 Week Triple P Self directed workbook
  Other Names: Triple P

SUMMARY:
The purpose of the study is to assess the characteristics of parents who enroll in parenting interventions and to assess the utility and efficacy of a self-directed Triple-P intervention for parents of children with a diagnosis of cancer. The study aims to recruit parent(s) or primary caregiver of children with a diagnosis of cancer.Participants will be parents of children aged between 3-10 years who have had a diagnosis of cancer for 6 months or more. Recruitment will take place nationally via cancer voluntary groups/charities and other relevant organisations. The project will be advertised through these organisations and their various media outlets such as newsletters and social media pages (e.g. Facebook). All data collection will take place online. Following completion of the initial survey, parents will have the option to opt in to a case series whereby 10 parents will have the opportunity to receive the Triple P Every parents self- directed workbook to complete over 10 weeks.

DETAILED DESCRIPTION:
The risk of developing cancer in childhood is around 1 in 500, with leukemia being the most common diagnosis. Eight out of ten children now survive for five years or more. Consequently, there is a growing need to support the survivors of cancer and their families post treatment, particularly in relation to psychosocial well-being. Despite some children achieving good psychological adjustment, there is an increasing recognition of emotional and behavioural problems in child cancer survivors. Children with cancer have shown significantly higher scores for hyperactivity/impulsivity, rule-breaking behaviours and aggressive behaviours when compared to healthy controls.

The Triple P - Positive Parenting Program is a successful treatment for emotional and behavioural difficulties designed to improve the quality of parenting advice available to parents through a multilevel system intervention. All forms of Triple P have shown to have moderate to large effects on parent reported child behaviours. More recently, self-directed Teen Triple P has been shown to be effective in reducing illness related conflict and behavioural problems in adolescents with type-1 diabetes.

There is emerging research addressing the predictors and barriers of parental enrolment and engagement to parenting programmes. Historically, factors studied in relation to participation and engagement have been limited in scope and often include socioeconomic disadvantage perceived need for help and rates of problem behaviours. Little is known about the parent factors associated with participation, particularly in a cancer population. Caring for a child with a chronic illness, such as cancer, typically causes significant and prolonged distress for parents. Whilst parental motivation has been shown to indicate engagement, stress and helplessness and increased negative life events have been linked to reduced efficacy and non- completion. However, there is a paucity of research indicating whether such factors affect enrolment for parents of children with a diagnosis of cancer.

A need for parenting information has been demonstrated by Williams et al who report that parents require information about parenting strategies particularly to manage challenging behaviours being exhibited by their child. In addition, at a local level, a survey undertaken with parents of children with a diagnosis of cancer attending the oncology service at the Royal Manchester Children's hospital has indicated a need for intervention, which is accessible and provides written support to parents for managing children's behavioural difficulties. The survey identified that 97% of parents believe parenting information should be given as a matter of routine following a child's diagnosis of cancer. Furthermore, parents reported a need for support with a range of behavioural difficulties, including tantrums and angry outbursts (43%). The purpose of the current study is to examine the predictors of parental enrollment to and pilot the efficacy of a self -directed version of the Triple P - Positive Parenting Program for parents of children with a diagnosis of cancer. Specifically the investigators aim to address whether a parent's experiences of their child's illness affects their ability to enroll to the study and whether Triple P is a suitably accessible intervention for parents of children with a diagnosis of cancer. Research suggests that interventions with minimal or no therapist or methods which promote self-regulation, such as written work books with self-directed exercises can be effectively employed to address child behaviour problems.To date, there have been no studies investigating self-directed measures to help parenting in the context of children with cancer. It is hoped the proposed project will determine the efficacy of this.

Aims:

To investigate the predictors of enrolment to a self-directed Triple P- Positive Parenting Program for parents of children with a diagnosis of cancer aged 3 to 10 years. Specifically, testing whether parents' perceived distress and emotional resource (as measured by the Parents Experience of Child Illness Questionnaire, PECI), psychosocial risk factors (as measured by the Family Background questionnaire; FBQ), parenting style (as measured by the parenting style questionnaire; PS), parental confidence (as measured by the parenting sense of competency questionnaire; PSOC), number of behavioural difficulties (measured by the Royal Marsden Hospital Pediatric Oncology quality of life measure; RMH-PQLQ), quality of life (measured by RMH-PQLQ) and cancer diagnosis predict enrolment to the intervention.

To assess the effectiveness of a self-directed Triple-P Positive Parenting Program in:

1. Improving quality of life as measured by the Royal Marsden Hospital Paediatric Oncology Quality of Life Questionnaire (RMH-PQLQ) (Primary outcome).
2. Reducing behavioural difficulties as measured by the Royal Marsden Hospital Paediatric Oncology Quality of Life Inventory (RMH-PQLQ) Life Questionnaire (Q's 47-67) (Secondary Outcome).
3. Promoting change in parenting style and feelings about being a parent as measured by the Parenting Scale (PS) and Parent self -confidence as measured by the Parenting Sense of Competence Questionnaire (PSOC) (Secondary Outcome).

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the trial.

  * Parent of a child with a diagnosis of cancer
  * Child has had cancer diagnosis for 6 months or more
  * Parent of a child aged between 3 and 10 years old
  * Parent can read unsupported
  * Parent and Child do not have a mental health diagnosis

Exclusion Criteria:

* Children between the ages of 0 to 2 years and 11 months and 11 years upwards

  * Children or parent has a mental health diagnosis
  * Parent unable to read without support or assistance
  * Parents of child who has been diagnosed with cancer for less than 6 months

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2016-01; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in Quality of life as measured by Royal Marsden Hospital Paediatric Oncology Quality of Life Questionnaire (RMH-PQLQ) | Week 1, Week 5, Week 10 and 1 month following completion.
  Improving quality of life

SECONDARY OUTCOMES:
Change in behavioural and emotional difficulties as measured by Royal Marsden Hospital Paediatric Oncology Quality of Life Inventory (RMH-PQLQ) Life Questionnaire | Week1, (baseline between 1-3 weeks), week 5, Week 10 and 1 month following completion
  Reducing behavioural and emotional difficulties (Q's 47-67) (Secondary Outcome).
Change in parenting style as measured by Parenting Scale (PS) | Week 1, Week 5, Week 10 and 1 month following completion.
  Promoting change in parenting style
Change in parental confidence as measured by Parenting Sense of Competence Questionnaire (PSOC) | Week 1, Week 5, Week 10 and 1 month following completion.
  Feelings about being a parent & confidence
Change in parents thoughts and feelings related to parenting a child with cancer as measured by Parent Experience of Childhood Illness questionnaire | Week 1, Week 5, Week 10 and 1 month following completion.
  thoughts and feelings related to parenting a child who has experienced a chronic illness or been diagnosed with another medical condition

CONTACTS AND LOCATIONS:
Overall Officials: Katie Swift, BSc, Principal Investigator — The University of Manchester
Locations (1):
- The University of Manchester, Manchester, United Kingdom